CLINICAL TRIAL: NCT03078829
Title: The Relation of GnRH Treatment to QTc Interval in Transgender Female Youth: A Time Series Study
Brief Title: The Relation of GnRH Treatment to QTc Interval in Transgender Females
Status: Terminated | Type: Observational
Why Stopped: investigator has left UCSF
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Stephen Rosenthal, Professor of Pediatrics, University of California, San Francisco
Other Study IDs: 16-19936
Record Dates: First submitted 2017-02-28; First posted 2017-03-13 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Gender Dysphoria
Keywords: gender identity; trans female; GnRH agonists; QTc interval
MeSH Terms: conditions — Gender Dysphoria | interventions — Therapeutics; histrelin; Injections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trans female adolescents: All transgender males to females youth in pubertal stage Tanner stage 4-5, starting GnRH agonist and estrogen treatment
  Interventions: Drug: Treatment with a GnRh agonists

INTERVENTIONS:
Drug: Treatment with a GnRh agonists — All patients will be treated with GnRH agonists
  Other Names: histrelin acetate 50mg (SUPPRELIN LA®); l(LUPRON DEPOT®) 30 mg for 3-month injections

SUMMARY:
Background: The QT interval of the electrocardiogram (ECG), corrected for heart rate (QTc), is a measure of the duration of ventricular repolarization and is a widely used marker of ventricular arrhythmia risk. Testosterone has a shortening effect on QTc length, and the QTc interval in males is shorter than in females after the onset of puberty. Transgender female adolescents are treated with GnRH agonists or spironolactone that suppress endogenous testosterone secretion and might increase the QT interval sufficiently to increase the risk for malignant ventricular arrhythmias. There are no current guidelines regarding monitoring QTc interval in transgender females undergoing GnRH agonist treatment.

Objective: To assess the effect of GnRH agonist treatment on QTc interval in transfemale youth.

Methods: A quasi-experimental time series study of transgender female adolescent, seen at UCSF Child and Adolescent Gender Center (CAGC) during 2017-2019.

Specific aims:

To assess the impact of GnRH agonist treatment on QTc interval length in transgender female adolescent

DETAILED DESCRIPTION:
This study is a quasi-experimental time series study, designed to examine the relation between GnRH agonist treatment for 6 months in transgender female youth and electrocardiographic change in QTc interval. Study subjects will be identified when visiting the UCSF Child and Adolescent Gender Center (CAGC). A baseline electrocardiogram (ECG) will be obtained in clinic before initiation of GnRH agonist treatment and at the 6 months follow up appointment.

Sampling scheme: Consecutive sample of transfemale patients presenting to UCSF CAGC (Child and Adolescent Gender Center) clinics meeting entry criteria, who consent to participate in this study

Recruitment strategy: The investigators will approach all transfemale patients with pubertal Tanner stage 4-5 who are ready to start GnRH agonist. From past experience in CAGC clinic, willingness of patients to participate in studies is high. The investigators plan that ECG will be available at clinic visits to further assist recruitment.

Retention strategy: Patients that are being treated in CAGC clinic are followed up every 3 months. Patients are very compliant with clinic visits as patients are eager to complete their transition. ECG is planned to be available at the 6 months clinic follow up visit.

Measurements: The investigators will assess QTc interval using a standard 12-lead ECG. The investigators will also measure serum levels of calcium, potassium and magnesium to rule out electrolyte abnormalities as a cause for QTc interval change, and testosterone, estradiol, LH and FSH levels to assess GnRH agonist effect. The laboratory analytes will be measured using standard procedures in place at the UCSF Laboratory, which is certified by Centers for Medicare and Medicaid Services, the California Department of Health Services, and the College of American Pathologists.

Outcome: A 12-lead ECG will be performed using standardized inspected equipment, at baseline and after 6 months of treatment. ECG reading and evaluation will be done by a board certified cardiologist. QT interval corrected for heart rate will be assessed using the Fridericia's correction (QTcF = QT/RR^0.33), which is currently preferred in accordance with the E14 ICH Guideline adopted by FDA and EMA in 2005. To minimize observer bias, the board certified cardiologist who will read the ECGs and determine QT interval length will be blinded to before or after status of GnRH agonist treatment.

Potential confounding variables: As this is a time series study with each participant serving as her own control, individual characteristics such as age, race and genetic factors are eliminated as confounding factors. Although this study has a within group design, typical disadvantages for such a research design, like learning effects, regression to the mean and secular trends do not seem to be relevant here. The investigators will need to monitor for factors that may change in the same participant over time and might act as a cofounders or mediators:

* Serum calcium, magnesium, and potassium levels
* BMI
* Starting other medications prolonging QT interval as: antihistamines, antiemetic or promotility drugs, azole antifungals, fluroquinolones, macrolides, antipsychotics, selective serotonin reuptake inhibitors.

Statistical issues

Analysis approach: A paired T test will be used for statistical analysis.

Data management plan: The investigators will use the Research Electronic Data Capture (REDCap) system to create forms (appendix 1) for entering study patients information. The investigators will use the REDCap installation, and will store the REDCap data on servers, located at the UCSF Minnesota Street data center. These servers are maintained behind a firewall in a secure server room; all servers are backed up regularly off-site.

Ethical considerations: This study involves obtaining an ECG, which has only minimal risk for the participants. Other information that is needed for this study, including blood tests and other measurements, is part of the regular clinical care in CAGC clinic. After the data is initially gathered and entered, it will be de-identified using a unique research identification number, to protect participant's privacy.

ELIGIBILITY:
Inclusion Criteria:

1. Transgender males to females in pubertal stage Tanner stage 4-5
2. starting GnRH agonist treatment

Exclusion Criteria:

1. Heart disease or arrhythmias at base line
2. Electrolyte abnormalities at baseline (abnormal serum levels of calcium, potassium or magnesium)
3. Failure to obtain informed consent from a parent or guarding or informed assent from a youth.

Min Age: 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female gender identity
Study Population: Transgender males to females meeting entrance criteria who receive care at UCSF CAGC (Child and Adolescent Gender Center) clinic in Mission Bay
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-08-21 (Actual); Study Completion 2017-08-21 (Actual)

PRIMARY OUTCOMES:
change in QTc Interval | 6 months
  A 12-lead ECG will be performed using standardized inspected equipment, at baseline and after 6 months of treatment, difference in milliseconds will be calculates

SECONDARY OUTCOMES:
QTc interval > 450 milliseconds | 6 months
  number of participants with QTc > 450 milliseconds at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No